CLINICAL TRIAL: NCT06690515
Title: Phase I/II, Open Label, Randomized, Safety and Immunogenicity Following DTwP-Hepatitis B-Hib-IPV Vaccine (Bio Farma) in Indonesian Infants
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Faculty of Medicine Universitas Padjadjaran (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hexa 010224
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Vaccine Adverse Reaction; Vaccine Reaction
MeSH Terms: interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula A (Experimental): 0,5 ml of DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula A injected three-dose regimen with 28 days interval between doses
  Interventions: Biological: DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula A
- DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula B (Experimental): 0,5 ml of DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula B injected three-dose regimen with 28 days interval between doses.
  Interventions: Biological: DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula B
- Registered DTwP-Hepatitis B-Hib Vaccine and IPV (Sinovac) ® (Active Comparator): 0,5 ml of DTwP-Hepatitis B-Hib Vaccine and IPV (Sinovac)® injected three-dose regimen with 28 days interval between doses.
  Interventions: Biological: Registered DTwP-Hepatitis B-Hib Vaccine and IPV (Sinovac)®

INTERVENTIONS:
Biological: DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula A — 0,5 ml DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula A injected three-dose regimen with 28 days interval between doses. Vaccine is injected intramuscularly in left anterolateral thigh.
  Arms: DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula A
Biological: DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula B — 0,5 ml injected of DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula B three-dose regimen with 28 days interval between doses. Injected intramuscularly in left anterolateral thigh.
  Arms: DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine Formula B
Biological: Registered DTwP-Hepatitis B-Hib Vaccine and IPV (Sinovac)® — The control group will receive 0,5 ml of Registered DTwP-Hepatitis B-Hib vaccine and 0,5 ml IPV (Sinovac)® injected in three-dose regimen with 28 days interval between doses. Registered DTwP-Hepatitis B-Hib Vaccine are injected intramuscularly into the left antero-lateral thigh region. IPV (Sinovac)® vaccine are injected intramuscularly into the right mid-lateral thigh region
  Arms: Registered DTwP-Hepatitis B-Hib Vaccine and IPV (Sinovac) ®

SUMMARY:
This trial is open label, comparative, randomized, phase I/II study, experimental, randomized, open-label, three arm parallel group study. The primary objective for phase I is to evaluate the safety of the DTwP-Hepatitis B-Hib-IPV (Bio Farma) vaccine within 7 days after each dose. The primary objective for phase II is to evaluate protectivity of DTwP-Hepatitis B-Hib-IPV (Bio Farma) vaccine.

DETAILED DESCRIPTION:
This trial is open label, comparative, randomized, phase I/II study. For phase I, approximately 75 subjects will be recruited and will seamlessly continue to phase II recruiting 390 subject, in total 465 subjects.

In this study, DTwP-Hepatitis B-Hib-IPV (Bio Farma) vaccine will be compared to an active control (Registered DTwP-Hepatitis B-Hib Vaccine and Registered Inactivated Polio Vaccine). There are 2 formulas of DTwP-Hepatitis B-Hib-IPV Vaccine which will be used in the study. The regimen of the vaccine is 0,5 ml injected three-dose regimen with 28 days interval between doses. On the other hand, the control group will receive 0,5 ml of Registered DTwP-Hepatitis B-Hib vaccine and 0,5 ml Inactivated Bio Farma vaccine injected in three-dose regimen with 28 days interval between doses.

The safety and immunogenicity result of the Phase I study will determine the continuation of the next phase clinical trial. Clinical trial of phase II can be conducted after safety observation within 28 days after the third dose in phase I. Three hundred and ninety (390) healthy subjects aged 6-11 weeks of age will be recruited in Phase II trial.

ELIGIBILITY:
Inclusion Criteria:

1. Infant 6-11 weeks of age.
2. Infant born after 37-42 weeks of pregnancy.
3. Infant weighing more than 2.5 kg at birth.
4. Father or mother, or legally acceptable representative properly informed about the study and signed the informed consent form.
5. Parents will commit themselves to comply with the indications of the investigators and with the schedule of the trial.

Exclusion Criteria:

1. Child concomitantly enrolled or scheduled to be enrolled in another trial.
2. Evolving moderate or severe illness, especially infectious diseases or fever (axillary temperature ≥37.5°C on Day 0).
3. Known history of allergy to any component of the vaccines.
4. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
5. Known history of congenital or acquired immunodeficiency (including HIV infection).
6. Child who has received in the previous 4 weeks of a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long term corticotherapy (> 2 weeks).
7. Other vaccination within the 7 days prior to inclusion with the exception of BCG and poliomyelitis.
8. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
9. Infant with a known history of diphtheria, tetanus, pertussis, Hib, hepatitis B infection.

Ages: 6 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 465 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safety of the DTwP-Hepatitis B-Hib-IPV (Bio Farma) vaccine within 7 days after each dose | From enrollment to 7 days after first dose
  Safety of the DTwP-Hepatitis B-Hib-IPV (Bio Farma) vaccine within 7 days after each dose
Phase II: Immunogenicity of DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine | From enrollment up to 28 days after third dose
  Protectivity of DTwP-Hepatitis B-Hib-IPV (Bio Farma) Vaccine

SECONDARY OUTCOMES:
Phase I: Safety of the vaccine within 28 days after last dose | From enrollment to 28 days after each dose
  Number and percentage of solicited and unsolicited adverse events within 28 days after each dose
Phase I: Safety of the vaccine within 6 months after last dose | From enrollment up to 6 months after the last dose
  Number and percentage of subjects with serious adverse events until 6 months after last dose
Phase I: Comparison of safety within 28 days after each dose between vaccines and active control | From enrollment to 28 days after each dose
  Comparison of number and percentage of subjects with adverse events between vaccine and control group within 28 days after each dose
Phase I: Comparison of safety until 6 months after last dose between vaccines and active control | From enrollment to 6 months after last dose
  Comparison of number and percentage of subjects with serious adverse events between vaccine and control group until 6 months after last dose
Phase I: Routine laboratory evaluation that probably related to the vaccination | From enrollment to 7 days after first dose
  Any deviation from routine laboratory evaluation that probably related to the dosing 7 days after first dose.
Phase I: Serological response to diphteria toxoid and tetanus toxoid | 28 days after the last dose immunization
  Serological response to diphtheria toxoid, tetanus toxoid: GMT, percentage of infants with titer ≥ 0.01 IU/ml, ≥ 0.1 IU/ml percentage of infants with increasing antibody titer ≥ 4 times and/or percentage of infants with transition of seronegative to seropositive.
Phase I: Serological response to the pertussis component (agglutinins) | 28 days after the last dose immunization
  GMT, percentage of infants with titer ≥ 40, ≥ 80 and ≥ 320 (1/dil.), percentage of infants with increasing antibody titer ≥ 4 times
Phase I: Geometric mean of anti-HbsAg | 28 days after the last dose immunization
  Percentage of infants with titer ≥ 10mIU/ml, percentage of infants with increasing antibody titer ≥ 4 times and/ or percentage of infants with transition of seronegative to seropositive.
Phase I: Serological response to Hib/PRP | 28 days after the last dose immunization
  GMT, percentage of infants with titer ≥ 1 μg /ml; ≥ 0.15 μg /ml percentage of infants with increasing antibody titer ≥ 4 times and/or percentage of infants with transition of seronegative to seropositive
Phase I: Serological response to polio type 1, 2, and 3 (humoral immunity) | 28 days after the last dose immunization
  GMT, percentage of infants with titer ≥ 8, percentage of infants with transition of seronegative to seropositive
Phase II: Serological response to diphtheria toxoid, tetanus toxoid | 28 days after the last dose immunization
  GMT, percentage of infants with titer ≥ 0.01 IU/ml, ≥ 0.1 IU/ml percentage of infants with increasing antibody titer ≥ 4 times and/or percentage of infants with transition of seronegative to seropositive
Phase II: Serological response to the pertussis component (agglutinins) | 28 days after the last dose immunization
  GMT, percentage of infants with titer ≥ 40, ≥ 80 and ≥ 320 (1/dil.), percentage of infants with increasing antibody titer ≥ 4 times
Phase II: Geometric mean of anti-HbsAg | 28 days after the last dose immunization
  percentage of infants with titer ≥ 10mIU/ml, percentage of infants with increasing antibody titer ≥ 4 times and/ or percentage of infants with transition of seronegative to seropositive.
Phase II: Serological response to Hib/PRP | 28 days after the last dose immunization
  GMT, percentage of infants with titer ≥ 1 μg /ml; ≥ 0.15 μg /ml percentage of infants with increasing antibody titer ≥ 4 times and/or percentage of infants with transition of seronegative to seropositive
Phase II: Serological response to polio type 1, 2, and 3 (humoral immunity) | 28 days after the last dose immunization
  GMT, percentage of infants with titer ≥ 8, percentage of infants with transition of seronegative to seropositive
Phase II: Safety of vaccine within 30 minutes after immunization | 30 minutes after immunization
  Local reaction and systemic events occurring within 30 minutes after immunization
Phase II: Safety of vaccine within 7 days after immunization | Within 7 days after immunization
  Local reaction and systemic events occurring within 7 days after immunization
Phase II: Safety of vaccine after 7 days to 28 days following the vaccination | From 7 days to 28 days following the vaccination
  Local reaction and systemic events occurring after the 7 days to 28 days following the vaccination

CONTACTS AND LOCATIONS:
Locations (3):
- Indonesia (3):
  - Garuda Primary Health Centre, Bandung, West Java
  - Ibrahim Adjie Priamry Health Centre, Bandung, West Java
  - Puter Primary Health Centre, Bandung, West Java

IPD SHARING:
Plan to Share IPD: No